CLINICAL TRIAL: NCT06610162
Title: Thermogenic Responses to Fasting and Overfeeding in Women: a Potential Mechanism Contributing to Postmenopausal Weight Gain
Brief Title: Thermogenenic Responses to Fasting and Overfeeding in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-1819
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: energy expenditure; adaptive thermogenesis; menopause
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This cross-sectional study will compare fasting and overfeeding effects on 24-hour EE and its components in pre- and postmenopausal women. We will study participants under three conditions in the room calorimeter: 1) eucaloric feeding (energy intake = EE); 2) acute, 24-hour fasting; and 3) acute, 24-hour overfeeding of a low-protein diet (i.e., 200% of energy requirements). Participants will complete the eucaloric study and then complete the overfeeding and fasting studies in random order. There will be a 1-4-week washout between conditions. Studies in premenopausal women will be performed during the mid-luteal phase (i.e., days 16-24) when both E2 and progesterone are elevated and, thus, when the potential hormonal effects are maximal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premenopausal women (Other)
  Interventions: Other: Eucalaloric feeding; Other: Acute Fasting; Other: Acute Overfeeding
- Postmenopausal women (Other)
  Interventions: Other: Eucalaloric feeding; Other: Acute Fasting; Other: Acute Overfeeding

INTERVENTIONS:
Other: Eucalaloric feeding — Participants will complete a 3-day diet run-in followed by an 24-hr in-patient visit in the room calorimeter. The energy content of the diet will be REE x 1.5 (30% fat, 55% carbohydrate, 15% protein). On the study day, will arrive at 7 AM and an IV catheter will be placed for blood draws, as described in the research plan. Participants will then enter the calorimeter at 0800, exit at 0700 the following day. Participants will be instructed to engage in primary sedentary behaviors. The energy content of the diet will be 1.3 x REE (~30% fat, 55% carbohydrate, and 15% protein at each meal). Breakfast will account for ~25% and lunch and dinner ~30-35% of total energy needs. Meals will be provided at 0900, 1300, and 1800, and a light snack will be provided at 2000.
Other: Acute Fasting — Participants will complete a 3d diet run-in followed by an 24h in-patient visit in the room calorimeter. The energy content of the diet will be REE x 1.5 (30% fat, 55% carbohydrate, 15% protein). On the study day, will arrive at 7 AM and an IV catheter will be placed for blood draws, as described in the research plan. Participants will then enter the calorimeter at 0800, exit at 0700 the following day. Participants will be instructed to engage in primary sedentary behaviors. Participants will complete a 24 hour fast while in the calorimeter. They will be permitted to consume non-caloric beverages (i.e., water, non-caloric and non-caffeinated soft drinks, caffeine-free tea, or decaffeinated coffee) but refrain from consuming any caloric food or beverages. Upon exiting the calorimeter, participants will be provided a meal from the University of Colorado Hospital Patient Kitchen.
Other: Acute Overfeeding — Participants will complete a 3d diet run-in followed by an 24h in-patient visit in the room calorimeter. The energy content of the diet will be REE x 1.5 (30% fat, 55% carbohydrate, 15% protein). On the study day, will arrive at 7 AM and an IV catheter will be placed for blood draws, as described in the research plan. Participants will then enter the calorimeter at 0800, exit at 0700 the following day. Participants will be instructed to engage in primary sedentary behaviors. The energy content of the diet will be 200% of energy requirements, based on EE measured during the eucaloric condition. Macronutrient intake will be 3% protein, 51% carbohydrate, and 46% fat. Breakfast will account for ~25% and lunch and dinner ~30-35% of total energy needs. Meals will be provided at 0900, 1300, and 1800, and a light snack will be provided at 2000.

SUMMARY:
This study plans to learn more about why menopause increases the risk of weight gain. During and after menopause, women are prone to increased weight gain. The weight gained is primarily body fat, particularly visceral or abdominal body fat. The excess gain in abdominal fat during menopause increases the risk of chronic metabolic diseases such as heart disease and diabetes. The increase in weight and body fat with menopause may be due to changes in metabolism related to the loss of estrogen. This study plans to compare how the metabolism of premenopausal and postmenopausal women responds to changes in energy intake. The investigators will compare the changes in energy expenditure that occur during a period of acute fasting (24 hours) and a period of consuming excess calories (overfeeding).

DETAILED DESCRIPTION:
This cross-sectional study will compare fasting and overfeeding effects on 24-hour EE and its components in pre- and postmenopausal women. The investigators will study participants under three conditions in the room calorimeter: 1) eucaloric feeding (energy intake = EE); 2) acute, 24-hour fasting; and 3) acute, 24-hour overfeeding of a low-protein diet (i.e., 200% of energy requirements). Participants will complete the eucaloric study and then complete the overfeeding and fasting studies in random order. For 3 days before each condition, the investigators will provide participants with an outpatient diet designed to meet free-living energy requirements (energy intake = 1.5 x REE) and stabilize macronutrient intake (15% protein, 30% fat, 55% carbohydrate). There will be a 1-4-week washout between conditions. Studies in premenopausal women will be performed during the mid-luteal phase (i.e., days 16-24) when both E2 and progesterone are elevated and, thus, when the potential hormonal effects are maximal.

Pre-study assessments - Once enrolled, participants will complete a pre-study assessment visit in the Clinical and Translational Research Center (CTRC) Outpatient Clinic, and the following assessments will be performed:

1. Resting energy expenditure (REE) - will be measured by indirect calorimetry using a metabolic cart coupled with a canopy system (Parvo Medics TrueOne) and used to estimate energy requirements during the eucaloric condition. REE in premenopausal women will be measured in the luteal phase. Participants will arrive after an overnight fast (&amp;gt;10 hours) between 7 and 9 AM. They will rest while remaining awake for 30 minutes in a temperature-controlled room (~70⁰ F). Oxygen uptake (VO2) and carbon dioxide production (VCO2) will be measured for 20 minutes and averaged over the final 15 minutes.
2. Body composition - Body composition will be measured using dual X-ray absorptiometry (DXA, Hologic Discovery, Waltham, MA).
3. Visceral adipose tissue (VAT) volume - VAT volume and subcutaneous fat area (SFA) will be measured using computed tomography (CT). An instrument dedicated to research activity will be used for all scans (Philips Gemini 64TF). Axial CT images will be obtained through the center of the L2-L3 and L4-L5 inter-vertebral disc spaces.

Study Procedures: Once the pre-screening assessments are completed, participants will be studied under three conditions in the room calorimeter.

Room calorimeter - 24-hour EE and substrate oxidation will be measured using whole-room indirect calorimetry.For three days before each calorimeter study, participants will be instructed to refrain from exercise and provided with all food to stabilize energy and macronutrient intake. The energy content of the diet will be REE x 1.5 (30% fat, 55% carbohydrate, 15% protein). Participants will arrive at 0700h after an overnight fast on the study day. An IV catheter will be inserted in an antecubital vein. Fasting blood samples will be obtained before breakfast and at the end of the 24-hour study and analyzed for leptin, FGF21, and thyroid hormones (TSH, total T3, free T4). The investigators will also measure sex steroids (E2, progesterone) in premenopausal women to confirm that participants are studied in the luteal phase.

Participants will enter the calorimeter at 0800, exit at 0700 the following day, and be instructed to engage in primary sedentary behaviors (e.g., reading, watching TV, using the computer). During the eucaloric and overfeeding studies, meals will be provided at 0900, 1300, and 1800, and a light snack will be provided at 2000. Participants will be instructed to turn out the lights and prepare for bed no later than 2300. Participants will record their time in bed during the first visit and be instructed to prepare for bed during the subsequent two visits. The CTRC nursing staff will confirm bedtimes. Participants will be awoken at 0600, and a 30-minute measurement of REE will be obtained.

Participants will be monitored during this time to ensure that they remain awake and motionless.

The energy content of the diet during the calorimeter study will vary according to the study condition:

During the eucaloric study visit, the energy content of the diet will be 1.3 x REE (~30% fat, 55% carbohydrate, and 15% protein at each meal). Breakfast will account for ~25% and lunch and dinner ~30-35% of total energy needs. During the overfeeding study, macronutrient intake will be 3% protein, 51% carbohydrate, and 46% fat. During the fasting study visit, participants will be permitted to consume non-caloric beverages (i.e., water, non-caloric and non-caffeinated soft drinks, caffeine-free tea, or decaffeinated coffee) but refrain from consuming any caloric food or beverages. Upon exiting the calorimeter, participants will be provided a meal from the University of Colorado Hospital Patient Kitchen.

Blood samples will also be obtained 30 minutes after each meal and snack during the eucaloric and overfeeding conditions; blood samples will be obtained at the same time during the fasting study. Blood samples during the calorimeter studies are obtained by asking participants to extend an arm through an airlock in the side of the calorimeter. The investigators will store these samples for potential future analysis (e.g., proteomics, metabolomics, and hunger and satiety hormones; see Future Directions). During each condition, a 24-hour urine sample will be collected and analyzed for urine nitrogen and urea nitrogen, which are needed to perform substrate oxidation calculations, as well as for 24-hour urinary catecholamines.

ELIGIBILITY:
Inclusion criteria for premenopausal women

* Age 18-45 years.
* Regular menses (no missed cycles in the previous year; cycle length 25-35 d).

Inclusion criteria for postmenopausal women

* No menses for at least 12 months
* Follicular stimulating hormone (FSH) ≥50 mIU/ml.
* Women who are within 2 years of the final menstrual period are preferred

The primary exclusion criteria are:

* Body mass index > 30 kg/m2
* Diabetes (fasting glucose >126 mg/dL).
* Thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) <0.5 or >5.0 mU/L
* Uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP >90 mmHg.

Additional exclusion criteria for postmenopausal women

* History or current use of estrogen-based hormonal therapy
* Women who have undergone surgical menopause.

Additional exclusion criteria for premenopausal women

* Current hormonal contraceptive use (past 6 mo.).
* Pregnant, lactating, or intention to become pregnant during the study period.

Participants who fail the thyroid and BP criteria will be considered for enrollment if they receive treatment for these conditions and are considered stable by their treating physician.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | 24 hours
  The number of calories burned over a set period of time

SECONDARY OUTCOMES:
Fibroblast growth factor 21 (FGF21) | 24 hours
  FGF21 is a hepatic cytokine that impacts energy expenditure
24 hour carbohydrate oxidation | 24 hours
  The amount of carbohydrate burned over 24 hours, measured in grams/24 hour
24 hour fat oxidation | 24 hours
  The amount of fat burned over 24 hours, measured in grams/24 hour
24 hour protein oxidation | 24 hours
  The amount of protein burned over 24 hours, measured in grams/24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The project will also produce data on the following: 24 h energy expenditure and substrate oxidation, body composition and visceral fat, laboratory screening measures, and blood and urine samples to measure changes in leptin, thyroid hormones, FGF21, catecholamines induced by each feeding condition. We will release summarized data and individual-level data that has been de-identified. 24-hour EE data will be summarized and released as minute-by-minute data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data that can be shared will be made available at the time of associated publication(s) (data underlying peer-reviewed journal articles). Data that can be shared will be available for three years after completion of the project or after the last relevant publication, whichever is later.
Access Criteria: We will share data in a generalist repository as controlled access. Our institutional IRB does not allow public (open access) sharing of individual participant data. Only qualified individuals within the scientific community who request access to validate and replicate published research findings or perform analyses aligning with the approved protocol will receive repository access. Data users also agree not to share or redistribute any data downloads. Any publications or presentations that use the shared dataset must appropriately acknowledge the data source, list authors, and cite the associated publications. The requestor's institutional IRB or equivalent body must approve the requested use of the data. Data requestors must sign a data transfer agreement outlining the agreement with the above conditions to gain access